CLINICAL TRIAL: NCT04641884
Title: Clinical, Biological and Histological Characteristics of Bullous Pemphigoid Induced by antiPD-1/PDL-1 Therapy: A National Retrospective Cohort Study
Brief Title: Bullous Pemphigoid Induced by antiPD-1/PDL-1 Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Bullous pemphigoid
Record Dates: First submitted 2020-04-09; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Bullous Pemphigoid; Immunotherapy; Programmed Cell Death Ligand 1
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not concerned — Not concerned

SUMMARY:
Immune checkpoint inhibitors (monoclonal antibodies targeting cytotoxic T lymphocyte-associated antigen-4 (CTLA-4), programmed cell death protein 1 (PD-1) or programmed death ligand 1 (PD- L1)) have revolutionized the treatment of many cancers. The widespread use of these treatments has triggered a new spectrum of immune related adverse events (irAE). Several cases of bullous pemphigoid (BP) triggered by antiPD-1/PDL-1 therapy have been reported, and their characteristics are currently poorly described in the literature. The investigators sought to collect the French cases of BP triggered by antiPD-1/PDL-1 therapy, and to describe their clinical, biological and histological characteristics.

In this national, retrospective, observational study, investigators included patients treated with antiPD-1/PDL-1 therapy, with a diagnosis of bullous pemphigoid occurring during treatment or up to 12 months after its discontinuation. Diagnosis of BP was made by the dermatologist and was based on the following criteria: compatible clinical presentation, compatible histopathology findings, positive direct immunofluorescence (DIF) studies, positive enzyme-linked immunosorbent assay BP180/enzyme-linked immunosorbent assay BP230.

DETAILED DESCRIPTION:
All members of French study Group on Autoimmune Bullous Skin Diseases and French group of Onco-dermatology were asked to report cases of bullous pemphigoid induced by antiPD-1/PDL-1 therapy from 2014 to 2019. In this retrospective, observational cohort study, investigators included patients treated with PD-1 or PD-L1 inhibitor, with a diagnosis of bullous pemphigoid occurring during treatment or up to 12 months after its discontinuation. Diagnosis of BP was made by the dermatologist and was based on the following criteria developed by the French Bullous Study Group : compatible clinical presentation (absence of atrophic scars, absence of mucosal involvement and absence of predominant bullous lesions on the neck and head), compatible histopathology findings (subepidermal blister on skin biopsy; and linear deposits of IgG and C3 along the basement-membrane zone), positive DIF studies, positive enzyme-linked immunosorbent assay BP180/enzyme-linked immunosorbent assay BP230. For each case, collected data were : sex, type of tumor, type of checkpoint inhibitor, age at the onset of the checkpoint inhibitor, time from the onset of BP compared to the onset of the PD-1 inhibitor, clinical presentation of BP, results of complementary exams (skin biopsies, enzyme-linked immunosorbent assay for BP180 and BP230 and indirect immunofluorescence studies if available); treatment of BP used, consequence on antiPD-1/PD-L1 therapy, course of the tumor, other irAEs. Overall tumor response was determined by the treating oncologist and classified using RECIST 1.1 (Response Evaluation Criteria in Solid Tumors).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients treated with PD-1 or PD-L1 inhibitor, with a diagnosis of bullous pemphigoid occurring during treatment or up to 12 months after its discontinuation.
* Diagnosis of the BP based on the following criteria: compatible clinical presentation (absence of atrophic scars, absence of mucosal involvement and absence of predominant bullous lesions on the neck and head), compatible histopathology findings (subepidermal blister on skin biopsy; and linear deposits of IgG and C3 along the basement-membrane zone)
* Positive direct immunofluorescence studies, positive enzyme-linked immunosorbent assay BP180/enzyme-linked immunosorbent assay BP230.

Exclusion Criteria:

* Pregnant women
* BP occurring more than 12 months after antiPD-1/PDL-1 therapy

Ages: 50 Years to 93 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Already descripted.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical situation of the patient features | One day
  Composite criteria consisting of the presence of prurit (Yes=0 or No=1). All the measure will give the rate of 0, the abnormal clinical situation
Clinical situation of the patient features | One day
  Composite criteria consisting of the presence of urticarial plaques (Yes=0 or No=1). All the measure will give the rate of 0, the abnormal clinical situation
Clinical situation of the patient features | One day
  Composite criteria consisting of the presence of the number of new blisters per day (less(=1) or more(=0) than 10). All the measure will give the rate of 0, the abnormal clinical situation.
Clinical situation of the patient features | One day
  Composite criteria consisting of eosinophil rate (more than the normal rate = 0 less =1). All the measure will give the rate of 0, the abnormal clinical situation.
Clinical situation of the patient features | One day
  Composite criteria consisting of the enzyme-linked immunosorbent assay for BP180 and BP230 presence =0 absence =1. All the measure will give the rate of 0, the abnormal clinical situation.

SECONDARY OUTCOMES:
BP treatments | One day
  Rate of corticosteroids, steroids-sparing drugs and other drugs
Cancer evolution | One day
  Rate of relapse remission death

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No